CLINICAL TRIAL: NCT01350596
Title: An Open Label, Randomized, 2x2 Crossover, Single Dose, Phase 4 Study To Determine The Pharmaceutical Bioequivalence Of Ibuprofen 50mg/Ml (Laboratórios Pfizer Ltda) Oral Suspension Versus Alivium ® 50mg/Ml (Mantecorp Indústria Química E Farmacêutica Ltda.) Oral Suspension, In Healthy Fasting Volunteers.
Brief Title: A Bioequivalence Study Of Ibuprofen 50mg/ml (laboratórios Pfizer Ltda) In The Oral Suspension Form.
Acronym: B4371004
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4371004; ICF: PBIO027/11
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Bioequivalence Study; Ibuprofen; Alivium
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference Drug (Active Comparator)
  Interventions: Drug: Alivium®
- Test Drug (Active Comparator)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Alivium® — 400mg of Ibuprofen equivalent to 8mL (50mg/mL) oral suspension of the Reference Drug
  Arms: Reference Drug
Drug: Ibuprofen — 400mg of Ibuprofen equivalent to 8mL (50mg/mL) oral suspension of the Test Drug
  Arms: Test Drug

SUMMARY:
An open label, randomized, 2x2 crossover, single dose, phase 4 study to determine the pharmaceutical bioequivalence of ibuprofen 50mg/ml (laboratórios pfizer ltda) oral suspension versus alivium ® 50mg/ml (mantecorp indústria química e farmacêutica ltda.) Oral suspension, in healthy fasting volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18 to 55 years old male or female subjects (Healthy is defined as absence of clinically relevant abnormalities identified by detailed medical history, complete physical examination, including blood pressure and heart rate measurements, 12-lead ECG and clinical laboratory tests).
* Volunteers' BMI - Body Mass Index must range from 18.5 to 24.9 (Dietary Guidelines for Americans), however, it can range to 15% of the upper limit (18.5 to 28.63) and total body weight >50kg.
* Signed and dated Informed Consent Form by the subject or legally acceptable representative. If subject and/or legally acceptable representative is unable to read the Informed Consent Form, an impartial witness may sign it.
* Subjects willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Evidence or history of hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic clinically significant disease (including drug allergies, except for seasonal allergies, asymptomatic, untreated at the time of dosing).
* Any condition that may possibly affect the drug absorption (e.g. gastrectomy).
* Volunteer presenting a drug abuse history [patients making use of marijuana and hashish will be excluded if they used these drugs in less than three months before the medical appointment, and volunteers who have used drugs such as cocaine, phencyclidine (PCP), crack and heroin, will be excluded if they used them in less than one year before the medical appointment].
* A positive drug test in urine (Methamphetamine, Opiate, Morphine, Marijuana, Cannabis, Amphetamine, Cocaine, Benzodiazepine, and Benzoylecgonine) or a positive test for alcohol before admission during periods 1 and 2.
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 serving = 150 mL of wine or 360 mL of beer or 45 mL of concentrated liquor) within 6 months from selection.
* If volunteer have participated in any experimental study or have taken any experimental drug within 6 months prior to baseline (ANVISA: RDC Resolution No. 34, June 3, 2008).
* 12-lead ECG demonstrating QTc> 450 msec at screening visit. If the QTc exceeds 450 msec, the ECG should be repeated twice and the average of the three QTc values should be used to determine patient's eligibility.
* Pregnant or breastfeeding women, women of childbearing potential who are unwilling or unable to use a non-hormonal acceptable contraception method, as described in this protocol, from at least 14 days before the first dose of study medication.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) before the first dose of study medication. Phytotherapic medicine and phytotherapic supplements should be discontinued 28 days before the first dose of study medication. With one exception, acetaminophen/paracetamol can be used at doses of 1 g/day. The limited use of nonprescription medications not considered as affecting the patient's safety or the general study results may be allowed on a case by case basis after sponsor's approval.
* Blood donation of approximately 500 mL within 3 months before dosage.
* Known hypersensitivity to Ibuprofen or chemically related compounds;
* Volunteers in whom acetylsalicylic acid, iodate and other Nonsteroidal anti-inflammatory drugs have induced asthma, rhinitis, urticaria, nasal polyps, angioedema, bronchospasm and other symptoms of allergic or anaphylactic reactions.
* Sensitivity History to heparin or heparin-induced thrombocytopenia.
* Unwillingness or inability to comply with the Lifestyle Guidelines described in this protocol.
* Other psychiatric or severe acute or clinically chronic condition or laboratory abnormality that may increase the risk associated with participation in the study or administration of investigational product, or which may interfere with the interpretation of study results and, in the opinion of the investigator, would make the patient inadequate to enter this study.
* A positive beta HCG test in women.
* If volunteer presents any condition that prevents his or her participation in the study, according to the opinion of the investigator.
* Volunteer with gastroduodenal ulcer, or previous or active gastrointestinal bleeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Test Drug and Reference Drug | Up to 16h
Area under the plasma concentration versus time curve from time zero to the last measurable concentration of Test Drug and Reference Drug (AUC(0-tlast)) | Up to 16h

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time zero to infinity of Test Drug and Reference Drug (AUC(0-inf)) | Up to 16h
Time to peak concentration of Test Drug and Reference Drug (Tmax) | Up to 16h
Half-life of Test Drug and Reference Drug (T1/2) | Up to 16h
Elimination rate constant (K el) | Up to 16h
Area under the curve from the time of dosing (AUC t/inf) extrapolated to infinity | Up to 16h

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Aparecida de Goiânia, Goiás, Brazil

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4371004&StudyName=A%20Bioequivalence%20Study%20Of%20Ibuprofen%2050mg/ml%20%28laborat%F3rios%20Pfizer%20Ltda%29%20In%20The%20Oral%20Suspension%20Form.